CLINICAL TRIAL: NCT03060122
Title: The Clinical Feasibility of Combining Cranial Electrotherapy Stimulation (CES Alpha-Stim) and Non-invasive Interactive Neurostimulation (InterX) for Optimized Rehabilitation Following Extremity Immobilization
Brief Title: Combining CES Alpha-Stim and InterX for Optimized Rehabilitation Following Extremity Immobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Benjamin Keizer, Pain Psychologist, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2017.026
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard Care (No Intervention): Patient's randomized to this arm will receive standard post operative/post immobilization physical therapy or occupational therapy rehabilitation care without the use of NIN or CES.
- NIN (InterX) and CES (Alpha-Stim) (Experimental): The Alpha-Stim Cranial Electrical Stimulation device applies a micro-current trans-cranially via electrodes attached to the ear.The electrical current is controlled through a handheld device. Standard treatment sessions lasting approximately 20-60 minutes.
  InterX Therapy (non-invasive) has been developed specifically for the treatment of acute and chronic pain. It is delivered on the skin of the involved area. The device will be applied by a trained therapist along the course of the dermatomes in the affected area. Electrical current is controlled through a handheld device. Standard treatment sessions last approx 20-45 min.
  The treatment will be delivered in conjunction with the rehab visit (physical or occupational therapy)
  Interventions: Device: NIN; Device: CES
- NIN (InterX) and sham CES (Active Comparator): The Alpha-Stim Cranial Electrical Stimulation device intensity will be preset and locked by the manufacturer at its lowest therapeutic dose at 100 mA, a sub-sensory level that serves as a sham treatment.
  InterX Therapy (non-invasive) has been developed specifically for the treatment of acute and chronic pain. It is delivered on the skin of the involved area. The device will be applied by a trained therapist along the course of the dermatomes in the affected area.Electrical current is controlled through a handheld device. Standard treatment sessions last approx 20-45 min.
  The treatment will be delivered in conjunction with the rehab visit (physical or occupational therapy)
  Interventions: Device: NIN; Device: Sham CES

INTERVENTIONS:
Device: NIN — The InterX device will be applied by a trained therapist along the course of the dermatomes in the affected area, paying special attention to the location of major cutaneous nerves ensuring optimal treatment points are identified and treated within the neurologically related area.
  Other Names: InterX
  Arms: NIN (InterX) and CES (Alpha-Stim); NIN (InterX) and sham CES
Device: Sham CES — The sham CES is identical to the regular device but ear clips will emit a dose at 100 mA, a sub-sensory level.
  Other Names: Alpha-Stim Sham
  Arms: NIN (InterX) and sham CES
Device: CES — Cranial Electrical Stimulation (CES) Alpha-Stim is a noninvasive medical treatment device that delivers a microcurrent (100 to 500 microamperes) via ear clip electrodes connected to a handheld device.
  Other Names: Alpha-Stim
  Arms: NIN (InterX) and CES (Alpha-Stim)

SUMMARY:
This study will be aimed at assessing the feasibility of a dual-device treatment prior to a rehabilitation session for an orthopaedic injury requiring immobilization, and its impact on improving outcomes and decreasing the risk for development of neuropathic pain. The investigators will evaluate the clinical feasibility and effectiveness of incorporating the Alpha-Stim and Inter-X treatment into a standard rehabilitation protocol to address risk factors associated with the development of neuropathic pain (i.e., pain, range of motion, and skin temperature) as well as its impact on reduced pain medication.

DETAILED DESCRIPTION:
Once patients provide consent and we have determined that they meet inclusion criteria the process will occur as follows:

1. Participants will be administered baseline demographic and standard medical history questionnaires, including information about prescription medication use. In addition, participants will fill out baseline self-report outcomes and be administered the (LANSS) Pain Scale. Range of motion and temperature will also be assessed during the initial session. Some of these measurements are standard of care and would be filled out by the participant even if the participant were not participating in the study.

Usual CARE The usual care aspect of this study is the delivery of the pain treatment (NIN and CES) as is commonly used at the Center for the Intrepid. The experimental aspect is the combined delivery of the treatment, and the use of sham treatment as a control. The treatment (NIN and CES) will be delivered in a pragmatic fashion, with treatment delivered in conjunction with rehab visits and lasting approximately 4-weeks total. Each session will last approximately 20-40 minutes long, and will most often be delivered in conjunction with their rehab visit (physical therapy or occupational therapy) that occurs anywhere from 1 to 3 times each week.

STRICTLY RESEARCH The experimental aspect of the study will be the comparison of combined treatment (NIN + CES), standard NIN with sham CES, to standard care alone. Before initiation of treatment participants will be randomized to either NIN + CES, NIN + Sham CES, or standard care only immediately after the immobilization device (cast, brace, etc) has been removed. Randomization with be performed with a random number gerator. All groups will continue with their own rehabilitation as indicated throughout the entire course of the study treatment, and beyond as indicated by their therapist. The investigators will keep track of rehab appointments and visits, but not control for them.

3. At the 1-month follow-up, all participants will fill out the same self-report outcome measures from baseline, to include prescription pain medication and be administered the LANSS pain scale. Range of motion and temperature will also be assessed.

4. At the 2 and 4-month follow-up the same assessments will again be administered. If the participant has completed formal therapy prior to the 2 and 4 month follow-up time points the participant will be asked to return to the clinic to complete these assessments. Participants may be contacted by telephone or email, if agreeable, to provide a reminder for the return appointment(s).

5. Outcomes will be compared between the three groups at each time point (i.e., initial, one month, two months, four months).

6. All participants will be followed out to 4 months.

Although every attempt will be made to collect data at these specific times, due to the variability of participant and clinic schedules, the actual timing of collection may vary (+/- 1 week) and some of the proposed measures may not be collected at all time points.

ELIGIBILITY:
Inclusion Criteria:

1. An orthopaedic/musculoskeletal postoperative injury that required cast or splint immobilization of the joint(s) to be treated of ≥ 2 weeks and available for treatment and are coming in for physical or occupational therapy
2. Between the age of 18 - 65 years
3. Read and speak English well enough to provide informed consent and follow study instructions

Exclusion Criteria:

1. Active infection, open sores, or open incisions (or anything that would inhibit the application of the stim) in the affected extremity.
2. Any contraindications to electrical stimulation including: any type of implanted demand type cardiac pacemakers, implanted defibrillators, or implanted functioning devices (i.e., insulin pump); active cancerous tissue or are undergoing chemotherapy; known pregnancy or breastfeeding or history of epilepsy or other seizures.
3. History of inflammatory skin diseases (psoriasis, dermatitis, etc.).
4. Contralateral extremity involvement resulting in less than normal range of motion, muscle strength, or daily pain greater than 1/10.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 4 months
  An 11-point verbalize NRS will be used to assess the subject's upper or lower extremity pain the day of each assessment as well as during therapy sessions. The 0 to 10 NPS has been found to be valid and reliable in many patient populations including the musculoskeletal population[37] and has been recommended for inclusion in the core NIH Toolbox for use with adults[38].

SECONDARY OUTCOMES:
Temperature | 4 months
  The temperature at three locations (different for upper and lower extremity) will be recorded with an infrared thermometer (Exergen DT-1001RS Infrared Dermal Thermometer with Remote Sensor, Exergen Corp, Watertown, Massachusetts) on both the involved and uninvolved extremities.
Range of Motion (ROM) | 4 months
  Active and/or passive ROM of the involved joints will be assessed using an electronic goniometer, and the reference of "normal" will be the non-involved limb. A measurement will be taken, but also the result will be dichotomously categorized as within 95% of opposite side - YES or NO.
Pain Medication | 4 months
  An 11-point verbalize NRS will be used to assess the subject's upper or lower extremity pain the day of each assessment as well as during therapy sessions. The 0 to 10 NPS has been found to be valid and reliable in many patient populations including the musculoskeletal population[37] and has been recommended for inclusion in the core NIH Toolbox for use with adults[38].
Global Rating of Change (GRC) | 4 months
  The GRC, a self-report instrument, assesses subjective perception of the efficacy of a particular treatment and the significance of that change [39]. A 15-point Likert type scale ranging from 1 (very great deal worse) to 15 (a very great deal better) and a 6-point Likert type scale ranging from 1 (a tiny bit important) to 6 (a very great important) will be used. The GRC is used to determine the minimal clinically important differences and will be used in this study to assess the participants' perceived magnitude of changes following the 30 minute combined NIN/CES treatment and again after each physical therapy or occupational therapy session for range of motion and pain.
The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale | 4 months
  The LANNS assessment helps identify whether or not a patient exhibits neuropathic pain. The instrument consists of five self-report and two clinician administered sensory function items that assess dynamic mechanical allodynia and altered pin-prick threshold (PPT). Weighted scores for the seven items are binary (yes or no) and summed, giving a total score between 0 and 24. In terms of diagnostic validity, during the validation study this assessment yielded a sensitivity of 85% and specificity of 80%[
National Institutes of Health Patient Reported Outcomes Measurement Information Systems (PROMIS) 29 | 4 months
  Emotional The PROMIS 29, a self-reported measure, assesses health-related quality of life (HRQOL) in seven domains (physical function, anxiety, depression, fatigue, sleep disturbance, social role satisfaction, pain interference, pain intensity). The instrument utilizes a 7-day recall period and consists of eight questions on a Likert-type scale, ranging from 1 to 5 , except for the pain intensity scale, which ranges from 0 to 10.
Lower Extremity Functional Scale(LEFS) | 4 months
  The LEFS, originally described by Binkley et al, provides global assessment of function related specifically to the lower extremities.[50] It is one self-report outcome measure that can capture adverse impact on function from multiple injuries or specific locations in the lower extremity. It consists of 20 questions total related to functional activities, each with a possible score ranging from 0 to 4, where 0 indicates that the activity cannot be performed at all and 4 indicates that the activity be performed with no limitations. The total maximum score is 80 points, indicating no limitations with any of the functional tasks. It has been shown to be valid, reliable, and responsive to change in various patient populations and in different body regions in the lower extremity (ankle, knee, and hip).[50-52]
Quick Disabilities of the Arm, Shoulder, and Hand (Quick DASH | 4 months
  The DASH is an 11-item self-report measure that assesses a subject's perceived ability to complete twenty-one upper extremity functional activities using a 5-point Likert scale. The cumulative Quick DASH score is scaled from 0 to 100, with higher scores indicating increased disability. The DASH is well tested and has been validated and found reliable in many different upper limb musculoskeletal disorders[45-48]. The Minimally Clinically Important Difference (MCID) for the Dash is 10.83 points, and for the QuickDash is 15.91 points.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Cancio, OTD, Study Director — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koltzenburg M. Neural mechanisms of cutaneous nociceptive pain. Clin J Pain. 2000 Sep;16(3 Suppl):S131-8. doi: 10.1097/00002508-200009001-00004. PMID 11014457
- [Background] Trescot AM, Helm S, Hansen H, Benyamin R, Glaser SE, Adlaka R, Patel S, Manchikanti L. Opioids in the management of chronic non-cancer pain: an update of American Society of the Interventional Pain Physicians' (ASIPP) Guidelines. Pain Physician. 2008 Mar;11(2 Suppl):S5-S62. PMID 18443640
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Webster BS, Verma SK, Gatchel RJ. Relationship between early opioid prescribing for acute occupational low back pain and disability duration, medical costs, subsequent surgery and late opioid use. Spine (Phila Pa 1976). 2007 Sep 1;32(19):2127-32. doi: 10.1097/BRS.0b013e318145a731. PMID 17762815
- [Background] Hortobagyi T, Dempsey L, Fraser D, Zheng D, Hamilton G, Lambert J, Dohm L. Changes in muscle strength, muscle fibre size and myofibrillar gene expression after immobilization and retraining in humans. J Physiol. 2000 Apr 1;524 Pt 1(Pt 1):293-304. doi: 10.1111/j.1469-7793.2000.00293.x. PMID 10747199
- [Background] Brandt KD. Response of joint structures to inactivity and to reloading after immobilization. Arthritis Rheum. 2003 Apr 15;49(2):267-71. doi: 10.1002/art.11009. No abstract available. PMID 12687522
- [Background] Nigam AK, Taylor DM, Valeyeva Z. Non-invasive interactive neurostimulation (InterX) reduces acute pain in patients following total knee replacement surgery: a randomised, controlled trial. J Orthop Surg Res. 2011 Aug 24;6:45. doi: 10.1186/1749-799X-6-45. PMID 21864362
- [Background] Gorodetskyi IG, Gorodnichenko AI, Tursin PS, Reshetnyak VK, Uskov ON. Non-invasive interactive neurostimulation in the post-operative recovery of patients with a trochanteric fracture of the femur. A randomised, controlled trial. J Bone Joint Surg Br. 2007 Nov;89(11):1488-94. doi: 10.1302/0301-620X.89B11.19352. PMID 17998187
- [Background] Gorodetskyi IG, Gorodnichenko AI, Tursin PS, Reshetnyak VK, Uskov ON. Use of noninvasive interactive neurostimulation to improve short-term recovery in patients with surgically repaired bimalleolar ankle fractures: a prospective, randomized clinical trial. J Foot Ankle Surg. 2010 Sep-Oct;49(5):432-7. doi: 10.1053/j.jfas.2010.05.007. Epub 2010 Aug 5. PMID 20688546
- [Background] Kirsch DL, Smith RB. The use of cranial electrotherapy stimulation in the management of chronic pain: A review. NeuroRehabilitation. 2000;14(2):85-94. PMID 11455071
- [Background] Smith RB, Tiberi A, Marshall J. The use of cranial electrotherapy stimulation in the treatment of closed-head-injured patients. Brain Inj. 1994 May-Jun;8(4):357-61. doi: 10.3109/02699059409150986. PMID 8081350
- [Background] Taylor AG, Anderson JG, Riedel SL, Lewis JE, Bourguignon C. A randomized, controlled, double-blind pilot study of the effects of cranial electrical stimulation on activity in brain pain processing regions in individuals with fibromyalgia. Explore (NY). 2013 Jan-Feb;9(1):32-40. doi: 10.1016/j.explore.2012.10.006. PMID 23294818
- [Background] Cook KF, Dunn W, Griffith JW, Morrison MT, Tanquary J, Sabata D, Victorson D, Carey LM, Macdermid JC, Dudgeon BJ, Gershon RC. Pain assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S49-53. doi: 10.1212/WNL.0b013e3182872e80. PMID 23479545